CLINICAL TRIAL: NCT01519219
Title: Assessment Of Liver Function in Patients Undergoing Hepatic Irradiation
Acronym: IC-Green
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2003.081; HUM00041352 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2011-09-23; First posted 2012-01-26 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Hepatic Irradiation
Keywords: hepatic irradiation; IC-GREEN

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hepatic Irradiation
  Interventions: Radiation: Hepatic Irradiation

INTERVENTIONS:
Radiation: Hepatic Irradiation — Patients who take part in this study are required to be scheduled for hepatic irradiation. For the purposes of this research, they will undergo IC-GREEN testing within 2 weeks prior to the start of radiation therapy

SUMMARY:
The goal of the trial is to assess the effect of radiation treatment on liver function as determined by indocyanine green extraction. The long term goal is to determine if individual assessment of liver function using the IC-Green method, either alone or in combination with other factors, will provide Radiation Induced Liver Disease (RILD) risk-estimates that are superior to the probabilistic method currently in use.

DETAILED DESCRIPTION:
Following intravenous injection, IC-GREEN is rapidly bound to plasma protein, of which albumin is the principle carrier (95%). IC-GREEN is taken up from the plasma almost exclusively by the hepatic parenchymal cells and is secreted entirely into the bile. It undergoes no significant extrahepatic or enterohepatic circulation. Simultaneous arterial and venous blood estimations have shown negligible renal, peripheral, lung or cerebro-spinal uptake of the dye. Therefore, the serum clearance rate (determined from serial serum concentration measurements at various times after intravenous injection) can serve as a useful index of liver function.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older, all gender, ethnicities and races
* Life expectancy of at least 12 weeks
* Zubrod performance status ≤ 2
* Baseline clinical assessments of liver function by complete history and physical examination
* Laboratory tests to be done within 6 weeks prior to start of radiation: CBC and platelets, liver function tests including SGOT, SGPT, Alkaline Phosphatase, and bilirubin, albumin, BUN, creatinine, PT/PTT, INR

Exclusion Criteria:

* Pregnant
* History of allergy or are sensitive to IC-Green, iodine or to radiographic media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who take part in this study are required to be scheduled for hepatic irradiation.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2004-11-24 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Baseline IC-GREEN elimination | 1 day
  Most subjects will have five IC-GREEN assessments. Graphical displays will be used to choose the form of a time-dependent model of IC-GREEN elimination. A mixed, possibly nonlinear model, with patient as random effect, will be fit to the data by the maximum likelihood principle. Profile confidence intervals for the parameters will be determined.

SECONDARY OUTCOMES:
Change in IC-green elimination after radiation therapy | 6 months
  Using model parameters, a cumulative distribution function for IC-GREEN elimination at each time point will be determined from the patients who do not contract RILD. This will result in a smooth estimate of the IC-GREEN assay results, from which lower normal bounds (at, for instance, the fifth percentile) can be established.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Lawrence, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States